CLINICAL TRIAL: NCT02398643
Title: Examine the Impact of Early Chronic Disease Management Education Following Hospital Discharge in Acute Exacerbation of COPD
Brief Title: Examine the Impact of Early Education on COPD Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB14-0504; AIHS-CRIO Project Grant (Other: Alberta Innovated Health Solutions (AIHS))
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Acute Exacerbation of COPD; COPD; Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Pulmonary Education (EPE) (Other): Patients randomized to EPE will receive focused education sessions by a Certified Respiratory Educator. Education sessions will start within two weeks of discharge from hospital.
  Interventions: Other: Pulmonary Education (PE)
- Usual Care (Other): Patients randomized to usual care will receive general education sessions by a Certified Respiratory Educator within the month of being discharged.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Pulmonary Education (PE) — Patients enrolled in PE will undergo focused education sessions following discharge from hospital.
  Arms: Early Pulmonary Education (EPE)
Other: Usual Care — Patients enrolled in usual care will receive general education sessions following discharge from hospital.
  Arms: Usual Care

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease primarily caused by smoking. COPD creates a tremendous burden to the healthcare system, as disease exacerbations result in frequent, prolonged hospitalizations. While originally considered a disease specific to the lung, data has shown that COPD is associated with substantial cardiovascular (CV) morbidity and mortality. Exacerbations of COPD requiring hospitalization result in marked patient deterioration, and heightened CV risk. The cause of the increased CV risk with stable COPD, and the exaggerated CV risk during exacerbations of the disease are unknown; however, it may be due to chronic inflammation which is exacerbated with a flare-up of the disease, and/or chronic inactivity which is similarly worsened with bed-rest during a hospitalization. Despite the impact of COPD on healthcare, there are relatively few studies examining how COPD inpatient care impacts on patient outcomes, inflammation and CV risk. Disease management programs, such as pulmonary rehabilitation and patient self-management education, are part of guideline therapy for COPD; however, these are not regularly implemented following a hospitalization, and how these interventions affect patient outcomes, behavior, physical activity, inflammation and CV risk have not been well studied. The proposed long-term project will examine how early referral to chronic disease management programs after hospital discharge, affect patient outcomes. This study will provide invaluable information about outpatient management for a disease which has a tremendous impact on healthcare.

DETAILED DESCRIPTION:
Purpose: To examine the impact of early pulmonary education (PE) following hospital discharge on QoL, pulmonary/CV outcomes and AECOPD hospitalizations.

Rationale: Studies have shown that education improves self-efficacy and QoL in COPD. Whether these improvements translate to increased exercise tolerance, physical activity, reduced CV risk and hospitalizations in patients recently discharged from hospital requires examination.

Hypothesis: Patients who receive early education will have improved QoL, pulmonary/CV outcomes, and less COPD hospitalizations in the 6 months following hospital discharge. Education will improve self efficacy, physical activity and QoL while reducing CV risk as compared to usual care.

Study Design & Subject Recruitment: In Calgary, patients discharged following an AECOPD hospitalization are referred to the Calgary COPD and Asthma Program (CCAP) where they are seen by a Certified Respiratory Educator 1-2 times within the month following discharge. For this study, patients will be recruited from the CCAP program and randomized into receiving usual care; general education sessions over the month following discharge, or the experimental arm; focused education following discharge from hospital. Patients found to have an acute cardiac injury, mobility issues or residence outside the greater Calgary area will be excluded. All education visits will be 1hr in length, and occur at a local outpatient clinic. The education will focus on patient self-management and will use Living Well with COPD supporting literature (www.livingwellwithcopd.com) designed to improve patient self-management and physical activity. All patients will be followed up 6 months after discharge and will be interviewed to assess disease status, management review and if there has been a history of recurrence or relapse of the AECOPD. Hospital admissions and length of stay will be obtained through electronic medical records as described above. Patient assessments will include: quality of life, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity (PWV), vascular function and systemic inflammation (TNF, MMP-2, IL-6 and CRP). All data will be collected before, immediately and 6 months after education. The control group will have the same data collected at the same scheduled time. See above for descriptions of methods.

Data Handling: Data will be entered onto a secure anonymized database.

Data Analysis: The influence of education on QoL, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity, vascular function and systemic inflammation will be evaluated using a multivariate mixed-model multivariate analysis of variance (MANOVA) with treatment (education vs. usual care) being a fixed between-group variable and time (pre, immediate post, 6months post) as a repeated variable.

Sample size: Based on previous work, a total sample size of 140 (70 in each group) will be sufficient to detect a clinically significant difference in QoL and a significant difference in hospital readmission rates. Based on outhe investigators r recent work, this sample could detect a 10% difference in PWV and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the pulmonary ward for an AECOPD will be offered participation into this arm of the study.

Exclusion Criteria:

* Patients found to have an acute cardiac injury during admission, mobility issues or residence outside the greater Calgary area will be excluded.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Vascular Function | Change in baseline vascular function post respiratory education and 6 months
  Peripheral arterial tone (PAT) and arterial stiffness will be used to assess vascular function.

SECONDARY OUTCOMES:
Inflammatory markers (IL-6) | Change in baseline IL-6 post respiratory education and 6 months
  IL-6: is an interleukin that acts as both a pro-inflammatory and anti-inflammatory cytokine
Inflammatory markers (TNF-alpha) | Change in baseline TNF-alpha post respiratory education and 6 months
  TNF-alpha
Inflammatory markers (MMP-2) | Change in baseline MMP-2 post respiratory education and 6 months
  MMP-2
Inflammatory markers (CRP) | Change in baseline CRP post respiratory education and 6 months
  CRP - -reactive protein is a non-specific serum marker of inflammation (range <8 is normal)
Quality of Life (QoL) | Change in baseline Quality of Life post respiratory education and 6 months
  COPD Assessment Tool (CAT) will be used to assess quality of life.
Quality of Life (QoL) | Change in baseline Quality of Life post respiratory education and 6 months
  St. George Respiratory Questionnaire (SGRQ) will be used to assess quality of life.
Quality of Life (QoL) | Change in baseline Quality of Life post respiratory education and 6 months
  COPD Self Efficacy Scale will be used to assess quality of life.
Dyspnea | Change in baseline dyspnea post respiratory education and 6 months
  Modified Medical Research Council Dyspnea Scale (MMRC) will be used to assess dyspnea (breathlessness)
Physical Activity | Change in baseline physical activity post respiratory education and 6 months
  Physical activity will be assessed by an accelerometer worn on the patients wrist or upper arm
Hospital Re-admissions | One year re-admission
  Re-admission rates for AECOPD will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Calgary, Calgary, Alberta, Canada